CLINICAL TRIAL: NCT00911365
Title: A Double-blind Placebo-controlled Randomized Clinical Trial of Autologous Mesenchymal Stem Cells in Patients With Multiple System Atrophy
Brief Title: Trial of Autologous Mesenchymal Stem Cells in Patients With Multiple System Atrophy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Philhyu Lee/Associate Professor, Severance Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4-2008-0137
Record Dates: First submitted 2009-05-26; First posted 2009-06-01 (Estimated); Last update posted 2011-08-04 (Estimated); Status verified 2011-07

CONDITIONS: Multiple System Atrophy
Keywords: voluntary participants; 75 years old or less
MeSH Terms: conditions — Multiple System Atrophy | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- normal saline (Placebo Comparator)
  Interventions: Biological: normal saline
- autologous mesenchymal stem cells (Experimental)
  Interventions: Biological: autologous mesenchymal stem cells

INTERVENTIONS:
Biological: autologous mesenchymal stem cells — 4*107 stem cell (100ml) Intra arterial infusion/ one time, then 4*107 stem cell(100ml)Intravenous infusion 3 times/monthly
  -> Total four times
  Arms: autologous mesenchymal stem cells
Biological: normal saline — saline
  Arms: normal saline

SUMMARY:
This study is based on positive results in open label trial of mesenchymal stem cells therapy in patients with Multiple System Atrophy (MSA).

ELIGIBILITY:
Inclusion Criteria:

* 75 Years Old or Less
* Multiple System Atrophy
* Voluntary Participants

Exclusion Criteria:

* Doubted dementia (MMSE < 24)
* Severe febrile condition
* Serum SGOT/SGPT three times above
* Malignant mass

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2008-05; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Scores on unified MSA rating scale | one month
  The statistical difference between scores before and after autologous mesenchymal stem cells treatment of unified MSA rating scale will be measured every month and every year using paired t-test.

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea